CLINICAL TRIAL: NCT02434146
Title: A Phase I/IIa Safety and Efficacy Study of Topical Phenylephrine Applied to Oral Mucosa in Bone Marrow Transplant Patients Receiving Cytoxan Plus Total Body Irradiation
Brief Title: Topical Phenylephrine Solution in Preventing Oral Mucosa in Bone Marrow Transplant Patients Receiving Cyclophosphamide and Total Body Radiation Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A company in China has decided to license the product
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UW14068; NCI-2015-00576 (Other: NCI Trial ID); 2015-0062 (Other: Institutional Review Board); A536700 (Other: UW Madison); SMPH\PEDIATRICS\PEDIATRICS (Other: UW Madison)
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2017-09

CONDITIONS: Neoplasm; Oral Mucosa; Transplant-Related Disorder
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (topical phenylephrine solution) (Experimental): Patients undergoing a cyclophosphamide and total body irradiation regimen receive topical phenylephrine solution via spray to the oral mucosa 15-20 minutes prior to each cyclophosphamide infusion, 25-30 minutes after the beginning of each cyclophosphamide infusion, and 15-20 minutes prior to each radiation treatment.
  Interventions: Drug: Topical Phenylephrine Solution

INTERVENTIONS:
Drug: Topical Phenylephrine Solution — Given topically via spray

SUMMARY:
This phase I/II trial studies the safety of topical phenylephrine solution and to see how well it works in preventing oral mucosa (mouth sores) in bone marrow transplant patients receiving cyclophosphamide and total body radiation therapy. Topical phenylephrine solution may prevent or lessen the severity of oral mucosa in patients receiving cyclophosphamide and total body radiation prior to undergoing a bone marrow transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of phenylephrine (topical phenylephrine solution) applied topically to the oral mucosa of bone marrow transplant patients treated with cyclophosphamide plus total body irradiation.

II. To determine the maximum tolerated dose (MTD) and recommended phase II dose of phenylephrine applied topically to the oral mucosa of bone marrow transplant patients treated with cyclophosphamide plus total body irradiation.

III. To evaluate the efficacy of phenylephrine applied topically to the oral mucosa in preventing and/or decreasing severity of oral mucositis in bone marrow transplant patients treated with cyclophosphamide plus total body irradiation.

OUTLINE: This is a phase I, dose-escalation study of topical phenylephrine solution followed by a phase II study.

Patients undergoing a cyclophosphamide and total body irradiation regimen receive topical phenylephrine solution via spray to the oral mucosa 15-20 minutes prior to each cyclophosphamide infusion, 25-30 minutes after the beginning of each cyclophosphamide infusion, and 15-20 minutes prior to each radiation treatment.

After completion of study treatment, patients are followed up weekly for 2 weeks and then at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Be planning to receive a conditioning regimen for stem cell transplant (SCT) consisting of cyclophosphamide and total body irradiation and must meet inclusion criteria for SCT which include:
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Patients must have no evidence of active infections at the time of transplantation
* Patients must be human immunodeficiency virus (HIV) non-reactive
* Females of childbearing potential must not be pregnant or breastfeeding on admission for conditioning for SCT and a pregnancy test will be required for all females of child-bearing potential
* Patients must have a pre-transplant multi-organ assessment with the following outcome:
* A resting ejection fraction of 50% or greater which increases with exercise as demonstrated by resting/exercise multigated acquisition (MUGA)
* A forced expiratory volume in one second (FEV1) of 60% or greater, a diffusion capacity of 50% or greater, and a oxygen partial pressure (PO2) of 80 mm mercury (Hg) or greater on pulmonary function testing
* A serum creatinine of equal or less than 2.0mg/Dl and a creatinine clearance of 50 mL/min or greater on 24 hour urine collection
* A total bilirubin of less than 2.5 mg/dL, unless these values are due to underlying hematologic malignancy
* An aspartate aminotransferase (AST) less than 2 times the upper limit of normal, unless these values are due to underlying hematologic malignancy
* Be able to tolerate topical application of phenylephrine to the oral mucosa
* All patients must sign a written informed consent

Exclusion Criteria:

* Open or unhealed wounds or ulcers in the oral cavity
* Current use or use within past two weeks of an monoamine oxidase inhibitor (MAOI)
* Primary or secondary tumor in the oral cavity
* Known allergy to phenylephrine
* Uncontrolled hypertension (defined as blood pressure in adults > 150/95)

  * Patients on anti-hypertensive medications are eligible if blood pressure is controlled
* Enrollment in any other mucositis prevention study from screening up to day 45 post-stem cell transplant
* Patients who are not eligible to receive SCT with cyclophosphamide and total body irradiation (TBI) conditioning because they do not meet transplant criteria are also not eligible for this phenylephrine study
* General exclusion criteria for transplant include:

  * Patients who have angina and/or congestive heart failure requiring treatment, or who have had a myocardial infarction within the past year
  * Patients who have had any complication that makes the risk of death during transplantation from non-malignant causes greater than the risk of relapse
  * Patients who have any active infection; if the infection is successfully treated, the patient may be reconsidered for transplantation at a later date
  * Patients with diabetes who are not controlled by medical management will be ineligible
  * Psychiatric illness requiring psychiatric counseling or medical intervention other than antidepressant medications may make an individual ineligible and will be considered on a case-by-case basis
  * Psychosocial assessment by the bone marrow transplant team may identify individuals for whom this form of therapy may be contraindicated; these decisions will be based upon estimated adequacy of patient support systems and prediction of patient's compliance with medications, required diagnostic procedures, and/or follow-up care
  * Patients who have an ECOG performance status of greater than 2
  * Patients who have decreased pulmonary function due to any disorder as demonstrated by a diffusion capacity of less than 50% of predicted, a FEV1 of less than 60% of predicted, or a PO2 of less than 80mmHg on pulmonary function testing
  * Patients who have a resting ejection fraction of less than 50%
  * Patients who have renal disease as demonstrated by a serum creatinine clearance of greater than 2.0 mg/dL and/or a creatinine clearance of less than 50 mL/min
  * Patients who are pregnant or breast feeding at the time of admission for conditioning
* Any mental or physical condition, in the opinion of the principal investigator (PI) or PI designee, which could interfere with the ability of the subject to understand or adhere to the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-05-14; Primary Completion 2016-04-27 (Actual); Study Completion 2017-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margo L. Hoover-Regan, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adult participants undergoing hematopoietic stem cell transplantation (SCT) who were to receive cyclophosphamide and TBI as the conditioning regimen. Participants were recruited from the University of Wisconsin Hospitals and Clinics between May 2015 and December 2015.
Period: Overall Study
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for the Oral Mucositis Severity
Description: The mucositis AUC will be estimated using the trapezoid method and summarized in terms of means, standard deviation, median and range. This analysis will be performed in both the extended cohort as well as in the historical controls.
Time Frame: Up to 3 months
Population: This study was closed prematurely due to decreased numbers of eligible subjects. The full target accrual number was not achieved, and AUC could not be estimated or analyzed.
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 0

2. Primary Outcome: Duration of Grade 2 Oral Mucositis
Description: If the grade 2 oral mucositis has not been resolved (to a grade < 2) by the last day of toxicity assessment, then the duration will be censored at the last date of toxicity assessment. Will be analyzed using the Kaplan-Meier method. The median duration of grade 2/grade 3 oral mucositis will be calculated and reported along with the corresponding 95% confidence interval. This analysis will be performed in both the extended cohort as well as in the historical controls.
Time Frame: Date of onset of grade 2 oral mucositis to the date of the resolution of the grade 2 oral mucositis, assessed up to 3 months
Population: This study was closed prematurely due to decreased numbers of eligible subjects. The full target accrual number was not achieved, and the median duration of oral mucositis could not be analyzed.
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 0

3. Primary Outcome: Duration of Grade 3 Oral Mucositis
Description: If the grade 3 oral mucositis has not been resolved (to a grade < 3) by the last day of toxicity assessment, then the duration will be censored at the last date of toxicity assessment. Will be analyzed using the Kaplan-Meier method. The median duration of grade 2/grade 3 oral mucositis will be calculated and reported along with the corresponding 95% confidence interval. This analysis will be performed in both the extended cohort as well as in the historical controls.
Time Frame: Date of onset of grade 3 oral mucositis to the date of resolution to grade < 3 oral mucositis, assessed up to 3 months
Population: as for outcome 2
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 0

4. Primary Outcome: Efficacy Response Rate for Preventing Oral Mucositis With Sufficient Accuracy
Description: If a patient experiences no higher than grade 2 oral mucositis, then s/he will be defined as a responder. If a patient experiences grade >= 3 oral mucositis, s/he will be defined as a non-responder. Specifically, the efficacy response rate will be estimated with a standard error of less than 15% and the length of the 95% confidence interval will be less than 50%. The efficacy response rate will be summarized in tabular format. The Wilson score method will be used to calculate the 95% confidence interval for the efficacy response rate for the extended cohort.
Time Frame: Up to 3 months
Population: This study was closed prematurely due to decreased numbers of eligible subjects. The full target accrual number was not achieved, and the efficacy response rate could not be estimated.
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 0

5. Primary Outcome: Incidence of Adverse Events, Graded According to the Common Terminology Criteria for Adverse Events Version 4.0
Description: Adverse events (AEs) will be presented in the summary tables by preferred term nested within the System Organ Class. Verbatim description, preferred term, and system organ class for all AEs will be contained in the patient data listings. All AEs occurring after enrollment and throughout the study period will be recorded. Each toxicity event will be assigned an attribution: unrelated, unlikely, possibly, probably, or definitely phenylephrine treatment related.
Time Frame: Up to 3 months
Population: This study was closed prematurely due to decreased numbers of eligible subjects. The full target accrual number was not achieved, and no study conclusions could be made.
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 0

6. Primary Outcome: Maximum Tolerated Dose (MTD), Defined as the Highest Dose Level of Phenylephrine Applied to the Oral Mucosa Where 0/3, 0/6, or 1/6 Patients Experience a Dose-limiting Toxicity
Description: Determine Maximum Tolerated Dose (MTD), the highest dose level of phenylephrine applied to the oral mucosa
Time Frame: During the conditioning regimen (radiation and cyclophosphamide treatment), which is anticipated to last 1 week.
Population: This study was closed prematurely due to decreased numbers of eligible subjects. The full target accrual number was not achieved, and MTD could not be determined.
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 0

7. Primary Outcome: Recommended Phase IIa Dose
Description: The dose of topical phenylephrine solution which will be recommended for a larger follow-up phase II efficacy study will be established after the dose cohort at the MTD has been expanded to a total of 12 patients.
Time Frame: During the conditioning regimen (radiation and cyclophosphamide treatment), which is anticipated to last 1 week.
Population: This study was closed prematurely due to decreased numbers of eligible subjects. The full target accrual number was not achieved, and the dose of topical phenylephrine solution for a larger follow-up phase II efficacy study could not be recommended.
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 0

8. Primary Outcome: Time to Onset of Grade 2 Oral Mucositis
Description: Will be analyzed using a parametric (one-parameter exponential) cure rate model. Will be performed in both the extended cohort as well as in the historical controls.
Time Frame: Time between the first date of radiation or cyclophosphamide treatment to the date of the onset of grade 2 oral mucositis, assessed up to 3 months
Population: This study was closed prematurely due to decreased numbers of eligible subjects. The full target accrual number was not achieved, and time to onset of grade 2 oral mucositis could not be analyzed.
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 0

9. Primary Outcome: Time to Onset of Grade 3 Oral Mucositis
Description: as for outcome 8
Time Frame: Time between the first date of radiation or cyclophosphamide treatment to the date of the onset of grade 3 oral mucositis, assessed up to 3 months
Population: This study was closed prematurely due to decreased numbers of eligible subjects. The full target accrual number was not achieved, and time to onset of grade 3 oral mucositis could not be analyzed.
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year.
Arm/Group | Supportive Care (Topical Phenylephrine Solution)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (Topical Phenylephrine Solution) (N=3)
Grade 2/3 mucositis (Gastrointestinal disorders) | 3

LIMITATIONS AND CAVEATS:
This study was closed prematurely due to decreased numbers of eligible subjects. The full target accrual number was not achieved, and no study conclusions could be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes